CLINICAL TRIAL: NCT04204499
Title: Analysis of Screen-detected Lung Cancers' Genomic Traits
Acronym: ASCENT
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 21919
Record Dates: First submitted 2019-12-11; First posted 2019-12-19 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
Keywords: Genomic signatures; Screen-detected cancer; Non-invasive biological and radiological parameters
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood collection will take place from consented patients at the time of anaesthetic induction pre-surgery, to include:
  * 4 x 10ml EDTA-Streck tubes for germline DNA/RNA and exploratory biomarker analyses
  * Tumour surplus to diagnostic and pathological requirements will be collected for whole exome sequencing and RNA profiling.
  * Archival Diagnostic FFPE blocks and slides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective, observational cohort study of patients undergoing surgical resection for low dose CT (LDCT) screen-detected lung cancer (detected through the SUMMIT study- ClinicalTrials.gov Identifier: NCT03934866/ lung screening programmes), in which translational research is a fundamental aspect.

DETAILED DESCRIPTION:
The ASCENT study seeks to examine the genomic signatures of screen-detected cancers, in order to categorise the biological behaviour of such lesions and correlate this against non-invasive biological and radiological parameters. From these data, the plan is to explore strategies to characterise LDCT-detected cancers through non-invasive means, which the researchers believe may prove key in mitigating potential screening-associated harms.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with confirmed lung cancer or probable lung cancer via LDCT screening.
2. Planned for, or completed primary surgical resection either for histologically confirmed lung cancer, or strongly suspected lung cancer.
3. Able to provide written informed consent (or verbal informed consent for participants consenting to retrospective diagnostic samples and data collection only).

Exclusion Criteria:

1. Treatment with neoadjuvant therapy for current lung malignancy as per local MDT treatment decision.
2. Known Active Human Immunodeficiency Virus (HIV), Hepatitis B virus, Hepatitis C Virus or Syphilis.

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screen detected lung cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 526 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Genomic exploratory research | 4 years
  Measuring the differences in chromosomal instability between fast- and slow-growing screen detected cancers, quantified by weighted genome integrity index (WGII) derived from whole exome sequencing (WES) data

CONTACTS AND LOCATIONS:
Overall Officials: Sam Janes, Principal Investigator — UCL
Locations (2):
- United Kingdom (2):
  - St Bart's Hospital, London
  - UCLH, London